CLINICAL TRIAL: NCT07160465
Title: Efficacy of a Smartphone Suicide Prevention App: A Single-blind, Randomized, Controlled Multicenter Study
Brief Title: Efficacy of a Smartphone Suicide Prevention App
Acronym: PreventS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Fondation FondaMental (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RECHMPL20_0072; 2024-A02330-47 (Other: ANSM)
Record Dates: First submitted 2025-07-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Suicide; Suicide Attempt
Keywords: Suicide; Suicide attempt
MeSH Terms: conditions — Suicide; Suicide, Attempted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 316 suicide attempters will benefit from the VigilanS program alone
- Interventional group (Experimental): 316 suicide attempters will benefit from the app emma in addition to Vigilans
  Interventions: Other: emma application

INTERVENTIONS:
Other: emma application — 1. Emma will allow the patient to spontaneously contact the VigilanS tele-clinician team via a simple and quick access (when the patient presses an ergonomic button with the VigilanS logo). He can also contact the National Service for Suicide Prevention (3114) or the French national emergency medical assistance service 24/7 (Samu).
  2. Experts of the field have defined response thresholds for targeted questions on suicide risk and emotional tension. If the patient's answers to these questions reach these thresholds, emma will automatically send a message to the nearest VigilanS center. In this case, a message will appear indicating to the patient that the nearest center will contact him as soon as possible, encourage him to review his strategies and resources available on the app's Home and direct him to the breathing space.
  3. Emma offers a Safety Plan module that will allow the patient to help him/her to put into practice what he/she will develop with the VigilanS team on a daily bas
  Arms: Interventional group

SUMMARY:
It is an interventional research, single-blind, randomized, controlled, multicenter, which involves only minimal risks and constraints.

Patients who attend to the emergency department following a SA (Suicidal Attempt) represent a key group of patients with an extremely high risk of suicide in the short term.

A main problem in suicide prevention is that the increase of symptoms and suicidal risk occurs most often in the natural environment of patients, away from the system of care. Thus, the main goal in allowing real-time risk detection would facilitate immediate interventions, probably the best way to prevent a suicidal act. Additionally, the evolution of the suicidal crisis is very variable from one subject to another, in duration and symptoms, and often very brief. In contrast, the tools used to assess suicidal thoughts have so far been limited to intermittent assessments separated by weeks, months or years, which does not take into account the fact that suicidal thoughts can be highly variable over a few hours and that suicide attempts can occur in response to a rapid increase in thoughts over periods as short as the day. Mobile health (mHealth) interventions are the only that can respond to these fluctuations over time.

We have developed the first French app (emma) for EMA (Ecological Momentary Assessment) , customised EMI (Ecological Momentary Intervention) and prediction of SB (suicidal behaviour). It was designed by integrating evidence-based suicide prevention strategies and recommendations for the development of apps in the field of mental health. Emma helps to strengthen the patient's connection to his healthcare system and social network. This study led to the development and subsequent deployment of VigilanS. VigilanS is a multi-regional innovative care program for the prevention of suicide relapse, which has been implemented in several emergencies departments in France.

Our hypothesis is that emma offers an unprecedented opportunity to increase the efficiency of VigilanS, both for patients, by restoring their social connections, and for health professionals, in a simple, fast and efficient way. Thanks to emma, the patient will have daily support adapted to his condition (emotion management modules, safety plan, calls in case of emergency). Emma will fit easily into the daily practice of health professionals (little binding, little time consuming) and will complete the range of care organized by VigilanS.

The main objective is to evaluate over a 6-months follow-up the efficacy of a smartphone app (emma) in addition to the VigilanS program on the prevention of a suicidal event (suicide, SA, hospitalization or emergency department for suicidal ideation) compared to the VigilanS program only.

DETAILED DESCRIPTION:
632 participants will be enrolled and randomized into 2 groups:

* Control group: 316 suicide attempters will benefit from the VigilanS program alone
* Interventional group: 316 suicide attempters will benefit from the emma app in addition to VigilanS

The duration of inclusions is 24 months. Each patient's participation period is 6 months and includes three visits (inclusion, at 3 and 6 months).

At each visit, a clinical assessment will be performed to characterise psychopathology and suicidal characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 or over
* Subject benefiting from the VigilanS program (after an admission to an emergency ward following a suicide attempt)
* Subject with his own smartphone (iOS/Androïd)
* Subject able to understand the nature, purpose and methodology of the study
* Subject must be covered by public health insurance
* Signed informed consent form

Exclusion Criteria:

* Subject unable to read or/and write French
* Planned longer stay outside the region that prevents compliance with the visit plan
* Being protected by the law (tutorship or curatorship)
* Being deprived of liberty by administrative decision
* Being in a period of exclusion compared to another protocol
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
occurrence of a suicidal event | within 6 months of inclusion.
  The primary endpoint is the occurrence of a suicidal event (suicide, SA, hospitalization, or emergency admission for suicidal ideation) within 6 months of inclusion.

SECONDARY OUTCOMES:
suicidal ideation | Up to 6 months after study inclusion
  Intensity and severity of suicidal ideation assessed with C-SSRS.
psychological pain | Up to 6 months after study inclusion
  Level of psychological pain assessed by a validated Likert scale.
Level of depression | Up to 6 months after study inclusion
  Level of depression assessed by QIDS
Loneliness | Up to 6 months after study inclusion
  Level of loneliness assessed by ESUL
social isolation | Up to 6 months after study inclusion
  Level of social isolation assessed by ISI
hopelessness | Up to 6 months after study inclusion
  Level of hopelessness assessed by BHS
Objective and subjective connections with the healthcare system | number of care visit until the end of the study, an average of 6 months
  Number of care visits for psychiatric problems and/or suicidal ideation
Objective and subjective connections with the healthcare system | Semi-directive interviews during the visit at 6 months
  Semi-directive interviews conducted with patients who agree to participate in the qualitative study, to explore experiences related to psychiatric care and suicidal ideation.
Objective and subjective experience of the app (interventionnal group only) | Up to 6 months after study inclusion
  Frequency of connection.
Objective and subjective experience of the app (interventionnal group only) | within 6 months of inclusion.
  Acceptability and satisfaction of patients assessed by monthly questionnaires in the app (Likert scales), by a self-questionnaire to be completed at the last visit (MARS scale) and, for 30 patients who agree to participate in the qualitative study, during the qualitative evaluation of the experience of emma users.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Montpellier, France